CLINICAL TRIAL: NCT04624516
Title: Effect of Self-structured Foot Exercise on the Incidence of Plantar Foot Diabetic Ulcer Recurrence Post Healing at Least One Month
Brief Title: Effect of Self-foot Exercise on the Incidence of Plantar Foot Diabetic Ulcer Recurrence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maria Suryani (Other)
Responsible Party: Sponsor-Investigator, Maria Suryani, PhD (candidate), St Elisabeth School Health Science
Organization: St Elisabeth School Health Science (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 4477112020
Record Dates: First submitted 2020-11-04; First posted 2020-11-10 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Diabetic Foot Ulcer; Diabetic Foot
Keywords: diabetic foot ulcer; diabetes melitus; ankle brachial index; diabetic neuropathy; exercise
MeSH Terms: conditions — Diabetic Foot; Diabetic Neuropathies; Motor Activity | interventions — Pliability

STUDY DESIGN:
Intervention Model Description: The exercise group was trained structured foot exercise and they did the exercise independently until 24 weeks or until the recurrence occurred The control group had usual care
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigator didn't know the groups. The assessor didn't know the groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The group received training in self-structured foot exercise and they were encouraged to do self-structure foot exercise 3 times a week. They received usual care
  Interventions: Other: self-structured foot exercise
- Control Group (No Intervention): the group received usual care

INTERVENTIONS:
Other: self-structured foot exercise — The exercise was done 3 times a week (15x/until they tired x 2set). The exercise used a flexible band with difference thickness (0,5 mm in the first 12 weeks and 0,65 mm in the second 12 weeks)
  Other Names: foot exercise; flexibility and resistance foot exercise
  Arms: Intervention group

SUMMARY:
The incidence of diabetic foot ulcer recurrence in one year can reach 35%. Plantar foot diabetic foot ulcer is the most frequently diabetic foot ulcer recurrence. The recurrence incidence can occur at least 14 days after the diabetic foot ulcer has healed. Physical activity and exercise are highly recommended for the prevention of diabetic foot ulcers. The study about the form of foot exercise to prevent a diabetic foot ulcer recurrence is still unclear. The major hypothesis was there is an effect of self-structured foot exercise on the plantar foot diabetic ulcer recurrences. The minor hypothesis was (1) The improvement of HbA1c, ABI, diabetic neuropathy examination score, callus, and walking speed can decrease the incidence of plantar foot diabetic ulcer (2) a self-structured foot exercise can decrease the incidence and the speed of incidence plantar doot diabetic ulcer recurrence. Participants were randomized into two groups: Exercise group (n=25) and control group (n=25). The exercise is the combination of flexibility and resistance exercise using a flexible band in 24 weeks. The incidence of plantar diabetic foot ulcers was monitored through the research process.

DETAILED DESCRIPTION:
1. Introduction

   Diabetic foot ulcers are a form of diabetes mellitus (DM) patients' foot problems, characterized by chronic wounds below the ankle, which can penetrate the skin to the dermis. Meta-analysis results in 2016 showed a global prevalence of diabetic foot ulcers of 6.3%. The incidence in Indonesia reaches 7.3 - 24%.

   Diabetic foot ulcers can result in amputation and even death in patients. The diabetic foot ulcer caused 85% of foot amputation cases and 2.48 times higher than for patients without ulcers in the next five years. Diabetic foot ulcers can provide a high economic burden for patients, families, and the country due to the healing period of diabetic foot ulcers and expensive maintenance costs.

   Healed diabetic foot ulcers can undergo recurrence. Approximately 26 -78% of all diabetic foot ulcer incidents are recurrence events. Prevalence of recurrence globally within one year, three years, and five years after diabetic foot ulcer healing is 40%, 60 %, and 65%. The prevalence of diabetic foot ulcer recurrence in Semarang, Indonesia country reaches 35.4 %. It indicates that post-cured diabetic foot ulcer patients have a very high risk for recurrence of diabetic foot ulcers.

   The high incidence of diabetic foot ulcer recurrence is closely related to the biological and behavioral factors of patients who have not been resolved, despite the healing. The previous studies explained that the risk factors for diabetic foot ulcer recurrence after recovery include the location of plantar ulcers, HbA1c > 7,5%, peripheral artery disease, peripheral neuropathy, the absence of callus, duration of ulcers, duration of DM, and limitations of foot musculoskeletal function.

   The International Working Group on Diabetic Foot (IWGDF) stress the importance of efforts to prevent the occurrence of diabetic foot ulcers.The act of performing foot exercises has not been a guideline in preventing diabetic foot ulcer recurrence, although exercise is highly recommended in all DM patients to prevent diabetic foot ulcers. The recent studies, limited to DM patients, showed that foot exercises designed for DM patients could increase joint range of motion, muscle strength, walking speed, ankle-brachial index (ABI) as well as lower HbA1c levels that are also risk factors for diabetic leg ulcer recursion. Self-structured foot exercises are a combination of foot resistance exercises using flexible bands and foot flexibility exercises performed independently by patients, with frequencies three times a week at home. The study aimed to prove the effect of self-structured foot exercise on plantar foot diabetic ulcer recurrence incidence after recovery of at least one month.
2. Methods

The study used a Randomised control trial (RCT) design. The study had approved by the ethics committee of the Faculty of Medicine, Diponegoro University. The participants of the study were patients with healed plantar foot diabetic ulcers who had been treated at two hospitals in Semarang Indonesia and had been selected consecutively. The study carried out random allocation using software into a control group and intervention group. The participants were directly supervised in the first three weeks and after that supervised using a mobile phone.

The demographics and characteristics related to diabetic foot ulcer history were collected. The changing of ABI, diabetic neuropathy examination score, HbA1c level, walking speed, and callus before and after intervention were collected also. The researchers took all of the data outcomes before the intervention, 12 and 24 weeks after foot exercises. The participants discontinued the intervention if they had recurrence before 24 weeks, and then data retrieval was carried out one last time. The time of recurrence incidence was recorded.

The analysis of data used a computer with SPSS. The researchers used the Shapiro Wilk normality test to see the distribution of numerical data. Homogeneity of respondents' characteristics and the changes difference in DNE, ABI, walking speed, and HbA1c levels were tested using independent T-tests, Man Whitney, Chi-Square, and Fisher tests. Changing in DNE, ABI, HbA1c levels, and walking speed were calculated by calculating the difference in the last data collection results with the preliminary data collection from respondents. The difference of calluses between two group after the intervention were tested also. Spearman's test was conducted to look at the effect of ABI improvements, DNE scores, HbA1c levels, and walking pace on the decrease in plantar foot diabetic ulcer recurrence. Recurrence data for participants who did not complete the outcome for 24 weeks were filled in according to the last condition found. Chi-square tests and relative risk (RR) calculations with 2x2 tables, Confidence Interval (CI) 95%, and significant levels of <5% were conducted to determine the effect of self-structured foot exercises on plantar foot diabetic ulcer recurrence incidence. A logistical regression multivariate test was conducted to look at the effect of self-structured foot exercises, on plantar foot diabetic ulcer recurrence with control on confounding variables. Cox's multivariate regression test was conducted to look at the effect of self-structured foot exercises on the timing of plantar foot diabetic ulcer recurrence events with control on confounding variables.

ELIGIBILITY:
Inclusion Criteria:

* signed an informed consent
* aged 40-60 years
* can walk within 5 meters
* recently healed plantar foot diabetic ulcer (1-12 months)

Exclusion Criteria:

* post amputation of right and left lower limb
* contracture of lower limb
* parkinson's
* osteomyelitis history
* paralysis

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2019-09-04 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
The number of plantar foot diabetic ulcer recurrence incidence | up to 12 weeks
  The number of plantar foot diabetic ulcer recurrence incidence after healing of the last plantar foot diabetic ulcer at least 1 month. The measurement of diabetic foot ulcer by the specialist doctor using Wagner diabetic ulcer classification
The number of plantar foot diabetic ulcer recurrence incidence | up to 24 weeks
  The number of plantar foot diabetic ulcer recurrence incidence after healing of the last plantar foot diabetic ulcer at least 1 month. The measurement of diabetic foot ulcer by the specialist doctor using Wagner diabetic ulcer classification
The time of plantar foot diabetic ulcer recurrence incidence | up to 24 weeks
  The time of plantar foot diabetic ulcer recurrence incidence is found after healing of the last plantar foot diabetic ulcer at least 1 month.

SECONDARY OUTCOMES:
change of ankle brachial index (ABI) | from the date of assignment until the date of plantar foot diabetic ulcer recurrence found, whichever comes first, assessed up to 12 weeks and 24 weeks
  ABI is the ratio of the systolic blood pressure measured at the ankle to that measured at the brachial artery using hand held dopler with an 8 Megahertz (MHz) doppler probe
change of HbA1c level | from the date of assignment until the date of plantar foot diabetic ulcer recurrence found, whichever comes first, assessed up to 12 weeks and 24 weeks
  HbA1c is Glycated haemoglobin that measured in the laboratory with national glycohemoglobin standardization program (NGSP)
change of diabetic neuropathy examination (DNE) score | from the date of assignment until the date of plantar foot diabetic ulcer recurrence found, whichever comes first, assessed up to 12 weeks and 24 weeks
  The accumulation score of the result measurement consists of eight item, two testing muscle strength, one a tendon reflex, and five sensation. The min-max score is 0-16. The score was determined by doing a physical examination.
change of walking speed | from the date of assignment until the date of plantar foot diabetic ulcer recurrence found, whichever comes first, assessed up to 12 weeks and 24 weeks
  Walking speed is the ratio between times measured while walking in second as fast as possible on a flat and flat trajectory at a certain distance. A track distance used in the study was 5 meter. The time of waking was measured using stopwatch
callus | from the date of assignment until the date of plantar foot diabetic ulcer recurrence found, whichever comes first, assessed up to 12 weeks and 24 weeks
  Callus is the thickness of the plantar skin area that can be determined by inspection

CONTACTS AND LOCATIONS:
Overall Officials: Maria Suryani, Study Chair — St. Elisabeth School Health Science (STIKES St Elisabeth Semarang)
Locations (1):
- St Elisabeth School Health Science (STIKES St. Elisabeth Semarang), Semarang, Central Java, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
the result of this study is available to cite another researchers
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: anytime
Access Criteria: mariahandoko22@gmail.com

REFERENCES:
- [Background] Pemayun TGD, Naibaho RM. Clinical profile and outcome of diabetic foot ulcer, a view from tertiary care hospital in Semarang, Indonesia. Diabet Foot Ankle. 2017 May 17;8(1):1312974. doi: 10.1080/2000625X.2017.1312974. eCollection 2017. PMID 28649296
- [Background] Soewondo P, Ferrario A, Tahapary DL. Challenges in diabetes management in Indonesia: a literature review. Global Health. 2013 Dec 3;9:63. doi: 10.1186/1744-8603-9-63. PMID 24299164
- [Background] Raghav A, Khan ZA, Labala RK, Ahmad J, Noor S, Mishra BK. Financial burden of diabetic foot ulcers to world: a progressive topic to discuss always. Ther Adv Endocrinol Metab. 2018 Jan;9(1):29-31. doi: 10.1177/2042018817744513. Epub 2017 Dec 12. PMID 29344337
- [Background] Khalifa WA. Risk factors for diabetic foot ulcer recurrence: A prospective 2-year follow-up study in Egypt. Foot (Edinb). 2018 Jun;35:11-15. doi: 10.1016/j.foot.2017.12.004. Epub 2017 Dec 28. PMID 29753996
- [Background] Schaper NC, Van Netten JJ, Apelqvist J, Lipsky BA, Bakker K; International Working Group on the Diabetic Foot (IWGDF). Prevention and management of foot problems in diabetes: A Summary Guidance for Daily Practice 2015, based on the IWGDF guidance documents. Diabetes Res Clin Pract. 2017 Feb;124:84-92. doi: 10.1016/j.diabres.2016.12.007. Epub 2016 Dec 18. PMID 28119194
- [Background] Bus SA, van Netten JJ, Lavery LA, Monteiro-Soares M, Rasmussen A, Jubiz Y, Price PE; International Working Group on the Diabetic Foot. IWGDF guidance on the prevention of foot ulcers in at-risk patients with diabetes. Diabetes Metab Res Rev. 2016 Jan;32 Suppl 1:16-24. doi: 10.1002/dmrr.2696. No abstract available. PMID 26334001
- [Background] Colberg SR, Sigal RJ, Yardley JE, Riddell MC, Dunstan DW, Dempsey PC, Horton ES, Castorino K, Tate DF. Physical Activity/Exercise and Diabetes: A Position Statement of the American Diabetes Association. Diabetes Care. 2016 Nov;39(11):2065-2079. doi: 10.2337/dc16-1728. No abstract available. PMID 27926890
- [Background] Diabetes Canada Clinical Practice Guidelines Expert Committee; Sigal RJ, Armstrong MJ, Bacon SL, Boule NG, Dasgupta K, Kenny GP, Riddell MC. Physical Activity and Diabetes. Can J Diabetes. 2018 Apr;42 Suppl 1:S54-S63. doi: 10.1016/j.jcjd.2017.10.008. No abstract available. PMID 29650112
- [Background] Jeffcoate WJ, Vileikyte L, Boyko EJ, Armstrong DG, Boulton AJM. Current Challenges and Opportunities in the Prevention and Management of Diabetic Foot Ulcers. Diabetes Care. 2018 Apr;41(4):645-652. doi: 10.2337/dc17-1836. PMID 29559450
- [Background] Peters EJ, Armstrong DG, Lavery LA. Risk factors for recurrent diabetic foot ulcers: site matters. Diabetes Care. 2007 Aug;30(8):2077-9. doi: 10.2337/dc07-0445. Epub 2007 May 16. No abstract available. PMID 17507693
- [Result] Armstrong DG, Boulton AJM, Bus SA. Diabetic Foot Ulcers and Their Recurrence. N Engl J Med. 2017 Jun 15;376(24):2367-2375. doi: 10.1056/NEJMra1615439. No abstract available. PMID 28614678
- [Result] Zhang P, Lu J, Jing Y, Tang S, Zhu D, Bi Y. Global epidemiology of diabetic foot ulceration: a systematic review and meta-analysis dagger. Ann Med. 2017 Mar;49(2):106-116. doi: 10.1080/07853890.2016.1231932. Epub 2016 Nov 3. PMID 27585063
- [Result] Walsh JW, Hoffstad OJ, Sullivan MO, Margolis DJ. Association of diabetic foot ulcer and death in a population-based cohort from the United Kingdom. Diabet Med. 2016 Nov;33(11):1493-1498. doi: 10.1111/dme.13054. Epub 2016 Jan 10. PMID 26666583
- [Result] Alavi A, Sibbald RG, Mayer D, Goodman L, Botros M, Armstrong DG, Woo K, Boeni T, Ayello EA, Kirsner RS. Diabetic foot ulcers: Part I. Pathophysiology and prevention. J Am Acad Dermatol. 2014 Jan;70(1):1.e1-18; quiz 19-20. doi: 10.1016/j.jaad.2013.06.055. PMID 24355275
- [Result] van Netten JJ, Price PE, Lavery LA, Monteiro-Soares M, Rasmussen A, Jubiz Y, Bus SA; International Working Group on the Diabetic Foot. Prevention of foot ulcers in the at-risk patient with diabetes: a systematic review. Diabetes Metab Res Rev. 2016 Jan;32 Suppl 1:84-98. doi: 10.1002/dmrr.2701. PMID 26340966
- [Result] Dubsky M, Jirkovska A, Bem R, Fejfarova V, Skibova J, Schaper NC, Lipsky BA. Risk factors for recurrence of diabetic foot ulcers: prospective follow-up analysis in the Eurodiale subgroup. Int Wound J. 2013 Oct;10(5):555-61. doi: 10.1111/j.1742-481X.2012.01022.x. Epub 2012 Jun 19. PMID 22712631
- [Result] Waaijman R, de Haart M, Arts ML, Wever D, Verlouw AJ, Nollet F, Bus SA. Risk factors for plantar foot ulcer recurrence in neuropathic diabetic patients. Diabetes Care. 2014 Jun;37(6):1697-705. doi: 10.2337/dc13-2470. Epub 2014 Apr 4. PMID 24705610
- [Result] Molines-Barroso RJ, Lazaro-Martinez JL, Beneit-Montesinos JV, Alvaro-Afonso FJ, Garcia-Morales E, Garcia-Alvarez Y. Predictors of Diabetic Foot Reulceration beneath the Hallux. J Diabetes Res. 2019 Jan 8;2019:9038171. doi: 10.1155/2019/9038171. eCollection 2019. PMID 30729135
- [Result] Wrobel JS, Najafi B. Diabetic foot biomechanics and gait dysfunction. J Diabetes Sci Technol. 2010 Jul 1;4(4):833-45. doi: 10.1177/193229681000400411. PMID 20663446
- [Result] Liao F, An R, Pu F, Burns S, Shen S, Jan YK. Effect of Exercise on Risk Factors of Diabetic Foot Ulcers: A Systematic Review and Meta-Analysis. Am J Phys Med Rehabil. 2019 Feb;98(2):103-116. doi: 10.1097/PHM.0000000000001002. PMID 30020090
- [Result] Matos M, Mendes R, Silva AB, Sousa N. Physical activity and exercise on diabetic foot related outcomes: A systematic review. Diabetes Res Clin Pract. 2018 May;139:81-90. doi: 10.1016/j.diabres.2018.02.020. Epub 2018 Feb 23. PMID 29477503
- [Result] Francia P, Gulisano M, Anichini R, Seghieri G. Diabetic foot and exercise therapy: step by step the role of rigid posture and biomechanics treatment. Curr Diabetes Rev. 2014 Mar;10(2):86-99. doi: 10.2174/1573399810666140507112536. PMID 24807636
- [Result] Francia P, Anichini R, De Bellis A, Seghieri G, Lazzeri R, Paternostro F, Gulisano M. Diabetic foot prevention: the role of exercise therapy in the treatment of limited joint mobility, muscle weakness and reduced gait speed. Ital J Anat Embryol. 2015;120(1):21-32. PMID 26738255
- [Result] Iunes DH, Rocha CB, Borges NC, Marcon CO, Pereira VM, Carvalho LC. Self-care associated with home exercises in patients with type 2 diabetes mellitus. PLoS One. 2014 Dec 5;9(12):e114151. doi: 10.1371/journal.pone.0114151. eCollection 2014. PMID 25479542
- [Result] Pound N, Chipchase S, Treece K, Game F, Jeffcoate W. Ulcer-free survival following management of foot ulcers in diabetes. Diabet Med. 2005 Oct;22(10):1306-9. doi: 10.1111/j.1464-5491.2005.01640.x. PMID 16176187
- [Result] Hedayatpour N, Falla D. Physiological and Neural Adaptations to Eccentric Exercise: Mechanisms and Considerations for Training. Biomed Res Int. 2015;2015:193741. doi: 10.1155/2015/193741. Epub 2015 Oct 12. PMID 26543850
- [Result] Cerrahoglu L, Kosan U, Sirin TC, Ulusoy A. Range of Motion and Plantar Pressure Evaluation for the Effects of Self-Care Foot Exercises on Diabetic Patients with and Without Neuropathy. J Am Podiatr Med Assoc. 2016 May;106(3):189-200. doi: 10.7547/14-095. PMID 27269974
- [Result] Kluding PM, Pasnoor M, Singh R, Jernigan S, Farmer K, Rucker J, Sharma NK, Wright DE. The effect of exercise on neuropathic symptoms, nerve function, and cutaneous innervation in people with diabetic peripheral neuropathy. J Diabetes Complications. 2012 Sep-Oct;26(5):424-9. doi: 10.1016/j.jdiacomp.2012.05.007. Epub 2012 Jun 18. PMID 22717465
- [Result] Sartor CD, Hasue RH, Cacciari LP, Butugan MK, Watari R, Passaro AC, Giacomozzi C, Sacco IC. Effects of strengthening, stretching and functional training on foot function in patients with diabetic neuropathy: results of a randomized controlled trial. BMC Musculoskelet Disord. 2014 Apr 27;15:137. doi: 10.1186/1471-2474-15-137. PMID 24767584
- [Result] Barone Gibbs B, Dobrosielski DA, Althouse AD, Stewart KJ. The effect of exercise training on ankle-brachial index in type 2 diabetes. Atherosclerosis. 2013 Sep;230(1):125-30. doi: 10.1016/j.atherosclerosis.2013.07.002. Epub 2013 Jul 14. PMID 23958264
- [Derived] Suryani M, Samekto W, Heri-Nugroho, Susanto H, Dwiantoro L. Effect of foot-ankle flexibility and resistance exercise in the secondary prevention of plantar foot diabetic ulcer. J Diabetes Complications. 2021 Sep;35(9):107968. doi: 10.1016/j.jdiacomp.2021.107968. Epub 2021 May 28. PMID 34187716